CLINICAL TRIAL: NCT00862979
Title: A Multi-center, Randomized, Open-label, Parallel Group Study Investigating the Renal Tolerability, Efficacy and Safety of a CNI-free Regimen (Everolimus and MPA) Versus a CNI-regimen With Everolimus in Heart Transplant Recipients
Brief Title: A Study Investigating the Renal Tolerability, Efficacy, and Safety of a CNI-free Versus a Standard Regimen in de Novo Heart Transplant (HTx) Recipients
Acronym: MANDELA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ADE14; 2007-002671-14
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Heart Transplantation
Keywords: Heart Transplantation; Cardiac Transplantation; CNI-sparing; renal function; CNI; Cyclosporine A; Everolimus; mycophenolic acid
MeSH Terms: interventions — Everolimus; Cyclosporine; Tacrolimus; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CNI-regimen (Active Comparator): CNI-regimen: cyclosporine A (CyA) or tacrolimus (TAC) with everolimus (EVR) with corticosteroids
  Interventions: Drug: Everolimus (EVR); Drug: cyclosporine A (CyA); Drug: tacrolimus (TAC); Drug: Corticosteroids
- CNI-free-regimen (Experimental): CNI-free regimen: everolimus (EVR) with MPA (either MMF or enteric coated mycophenolate sodium (EC-MPS)) and corticosteroids
  Interventions: Drug: Everolimus (EVR); Drug: cyclosporine A (CyA); Drug: tacrolimus (TAC); Drug: Enteric coated mycophenolate sodium (EC-MPS); Drug: mycophenolate mofetil (MMF); Drug: Corticosteroids

INTERVENTIONS:
Drug: Everolimus (EVR) — Everolimus 0.25mg, 0.75mg or 1.0mg based on blood levels (5-10 ng/mL)
  Other Names: Certican, RAD001
Drug: cyclosporine A (CyA) — 10 mg, 25 mg, 50 mg or 100 mg capsule according to blood levels for CNI-regimen group. For CNI-free-regimen dispense on month 6 to 9 only
  Other Names: Sandimmun Optoral
Drug: tacrolimus (TAC) — 0.5 mg, 1 mg, or 5 mg capsule given according to blood levels for CNI-regimen. For CNI-free-regimen give on month 6 to 9 only
  Other Names: Prograf
Drug: Enteric coated mycophenolate sodium (EC-MPS) — 180 mg or 360 mg tablet dosed 1440-2280 mg per day
  Other Names: Myfortic
  Arms: CNI-free-regimen
Drug: mycophenolate mofetil (MMF) — 250 mg or 500 mg tablets with a dose of 1500-3000 mg per day
  Other Names: CellCept
  Arms: CNI-free-regimen
Drug: Corticosteroids — according to local standard: 0.05-0.3 mg/kg of prednisolone or equivalent

SUMMARY:
This study will assess whether a calcineurin inhibitor (CNI)-free regimen with everolimus and mycophenolic acid is associated with a better renal outcome as compared to the standard regimen containing cyclosporine A (which belongs to the class of CNIs) and everolimus; while both treatments are expected to be comparable with respect to efficacy.

DETAILED DESCRIPTION:
This study will assess whether a calcineurin inhibitor (CNI)-free regimen with everolimus and mycophenolic acid is associated with a better renal outcome as compared to the standard regimen containing cyclosporine A (which belongs to the class of CNIs) and everolimus; while both treatments are expected to be comparable with respect to efficacy.

ELIGIBILITY:
Inclusion criteria:

* Heart transplantation, 3 months prior to enrollment
* Patients have to receive an immunosuppressive regimen with Sandimmun® Optoral, Certican® and corticosteroids
* Sufficient graft function
* Sufficient renal function
* Females capable of becoming pregnant must have a negative serum pregnancy test within 7 days prior to or at baseline, and are required to practice an approved method of birth control for the duration of the study and for a period of 6 weeks following discontinuation of study medication, even where there has been a history of infertility

Exclusion criteria:

* Multi-organ recipients, re-transplantation, or previous transplant with any other organ.
* Patients who are recipients of A-B-O incompatible transplants
* Cold ischemia time >6 hours
* Historical or current peak PRA of > 25% at time of transplantation
* Already existing antibodies against the HLA-type of the receiving transplant Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-02-24 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Germany (9):
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Regensburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 232 patients were screened, of these , 193 patients were included in safety set which included 31 non-randomized and 162 randomized. Of these, 145 patients were treated with study medication and had at least 1 post-baseline assessment of the primary outcome variable and included in the Full Analysis Set FAS.
Period: Overall Study
Arm/Group | CNI-regimen | CNI-free-regimen
Started | 84 | 78
Full Analysis Set (FAS) | 74 | 71
Completed | 76 | 71
Not Completed | 8 | 7
Not completed — Adverse Event | 6 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Patient withdrew consent | 2 | 1
Not completed — Administrative problems | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set FAS- 145 patients were treated with study medication and had at least 1 post-baseline assessment of the primary outcome variable
Groups:
- Total: Total of all reporting groups
Arm/Group | CNI-regimen | CNI-free-regimen | Total
Number analyzed (Participants) | 74 | 71 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Full Analysis Set FAS- 145 patients were treated with study medication and had at least 1 post-baseline assessment of the primary outcome variable
  years | 52.7 (9.7) | 50.3 (9.8) | 51.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full Analysis Set FAS- 145 patients were treated with study medication and had at least 1 post-baseline assessment of the primary outcome variable
  Participants
    Female | 9 | 12 | 21
    Male | 65 | 59 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Full Analysis Set FAS- 145 patients were treated with study medication and had at least 1 post-baseline assessment of the primary outcome variable
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 74 | 71 | 145
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Calculated Glomerular Filtration Rate (cGFR) Using Modification of Diet in Renal Disease (MDRD) Formula at Month 18
Description: Calculated Glomerular Filtration Rate (cGFR) Using Modification of Diet in Renal Disease (MDRD) Formula at Month 18 cGFR (in mL/min/1.73 m2) = 186.3*(C-1.154)*(A-0.203)*G*R where C = the serum concentration of creatinine (mg/dL), A = age (years), G = 0.742 when gender is female, otherwise G = 1, R = 1.21 when race is black, otherwise R = 1.
Time Frame: Month 18
Population: Full Analysis Set-Last observation carried forward (FAS-LOCF)- 145 patients were treated with study medication and had at least 1 post-baseline assessment of the primary outcome variable but for this analysis only participants that had values at Month 18 were analyzed
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | CNI-regimen | CNI-free-regimen
Number analyzed (Participants) | 69 | 65
mL/min | 54.2 (17.9) | 66.9 (23.0)
Statistical Analysis 1: Comparison: CNI-regimen vs CNI-free-regimen; Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Net) = -11.3, 95% CI 2-sided [-16.5 to -6.1]

2. Secondary Outcome: Occurrence of Treatment Failures From Month 6 to 9 and Month 9 to 18
Description: Treatment failure was defined as composite endpoint of biopsy proven acute rejection of ISHLT 1990 grade ≥ 3A resp. ISHLT 2004 grade ≥ 2R, acute rejection episodes associated with hemodynamic compromise, graft loss / re-transplant, death, loss to follow up (at least one condition must be present). If participant had an occurrence in each period it was counted for each period.
Time Frame: Month 6 to Month 9; Month 9 to Month 18
Population: as for baseline characteristics
Measure: Number; unit: Occurences
Arm/Group | CNI-regimen | CNI-free-regimen
Number analyzed (Participants) | 74 | 74
Occurences
  Month 6 to Month 9 Treatment failure - all reasons | 1 | 4
  Month 9 to Month 18 Treatment failure-all reasons | 3 | 15
Statistical Analysis 1: Comparison: CNI-regimen vs CNI-free-regimen; Month 6 to Month 9; Test type: Other — difference; p = 0.203, Fisher Exact
Statistical Analysis 2: Comparison: CNI-regimen vs CNI-free-regimen; Month 9 to Month 18; Test type: Other — difference; p = 0.002, Fisher Exact

3. Secondary Outcome: Occurrence of Major Cardiac Events (MACE) From Month 6 to 18
Description: Major cardiac events (MACE) was defined as one of the following: any death, myocardial infarction, coronary artery bypass grafting
Time Frame: Month 6 to Month 18
Population: as for baseline characteristics
Measure: Number; unit: Occurences
Arm/Group | CNI-regimen | CNI-free-regimen
Number analyzed (Participants) | 74 | 71
Occurences
  Myocardial infarction | 1 | 0
  Death | 0 | 1

4. Secondary Outcome: Calculated Glomerular Filtration Rate (cGFR) According to Cockcroft-Gault at Month 12 and 18
Description: Calculated Glomerular Filtration Rate (cGFR) according to Cockcroft-Gault at Month 12 and 18. For men: GFR=(140-Age) x Body weight (kg) / 72 x Serum Creatinine (mg/dl) For women: GFR=0.85 (140 -Age) x Body weight(kg)/ 72 x Serum Creatinine (mg/dl)
Time Frame: Month 12 and 18
Population: Full Analysis Set-Last observation carried forward (FAS-LOCF)- 145 patients were treated with study medication and had at least 1 post-baseline assessment of the primary outcome variable but for this analysis only participants that had values at Month 12 & 18 were analyzed
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | CNI-regimen | CNI-free-regimen
Number analyzed (Participants) | 74 | 71
mL/min
  Month 12: number analyzed (Participants) | 68 | 62
  Month 12 | 54.2 (19.7) | 69.8 (23.4)
  Month 18: number analyzed (Participants) | 69 | 65
  Month 18 | 54.2 (17.9) | 66.9 (23.00)
Statistical Analysis 1: Comparison: CNI-regimen vs CNI-free-regimen; Month 12; Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Final Values) = -14.0, 95% CI 2-sided [-19.6 to -8.3]
Statistical Analysis 2: Comparison: CNI-regimen vs CNI-free-regimen; Month 18; Test type: Superiority; p < .0001, ANCOVA; Mean Difference (Final Values) = -11.3, 95% CI 2-sided [-16.5 to -6.1]

5. Secondary Outcome: Serum Creatinine at Month 6, 8, 9, 10 12 and 18
Description: Serum Creatinine is an indicator of renal function measured in the blood
Time Frame: Month 6, 8, 9, 10 12 and 18
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | CNI-regimen | CNI-free-regimen
Number analyzed (Participants) | 74 | 71
μmol/L
  Month 6 | 1.53 (0.49) | 1.49 (0.51)
  Month 8: number analyzed (Participants) | 73 | 70
  Month 8 | 1.44 (0.41) | 1.27 (0.35)
  Month 9: number analyzed (Participants) | 74 | 70
  Month 9 | 1.58 (0.75) | 1.24 (0.32)
  Month 10: number analyzed (Participants) | 74 | 70
  Month 10 | 1.53 (0.53) | 1.20 (0.30)
  Month 12: number analyzed (Participants) | 74 | 70
  Month 12 | 1.53 (0.52) | 1.22 (0.33)
  Month 18 | 1.50 (0.50) | 1.27 (0.44)

6. Secondary Outcome: Reciprocal Creatinine Slope Between Month 6 and Month 18
Description: Reciprocal Creatinine Slope is an indication of renal function over time with a higher slope value indicating an improvement in renal function.
Time Frame: Between Month 6 and Month 18
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: 1/(μmol/L)/(hour)
Arm/Group | CNI-regimen | CNI-free-regimen
Number analyzed (Participants) | 74 | 71
1/(μmol/L)/(hour) | 0.045 (0.364) | 0.403 (1.863)
Statistical Analysis 1: Comparison: CNI-regimen vs CNI-free-regimen; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Groups:
- CNI-free-regimen: CNI-free regimen: MPA (either MMF or enteric coated mycophenolate sodium (EC-MPS)) and everolimus and corticosteroids; On month 6 to 9 only: Cyclosporin A or tacrolimus
Arm/Group | CNI-regimen | CNI-free-regimen
All-Cause Mortality (participants affected / at risk) | 0/84 | 1/78
Serious Adverse Events (participants affected / at risk) | 40/84 | 29/78
Other Adverse Events (participants affected / at risk) | 74/84 | 65/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CNI-regimen (N=84) | CNI-free-regimen (N=78)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 3
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 1
HYPERTHYROIDISM (Endocrine disorders) | 1 | 0
EYE PAIN (Eye disorders) | 0 | 1
GLAUCOMA (Eye disorders) | 0 | 1
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 | 0
APHTHOUS ULCER (Gastrointestinal disorders) | 0 | 1
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 2
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 1
CHEST PAIN (General disorders) | 1 | 0
CHILLS (General disorders) | 0 | 1
FATIGUE (General disorders) | 0 | 1
OEDEMA (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PYREXIA (General disorders) | 0 | 2
STENOSIS (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 2 | 0
HEART TRANSPLANT REJECTION (Immune system disorders) | 3 | 7
ANAL ABSCESS (Infections and infestations) | 0 | 1
ASPERGILLOMA (Infections and infestations) | 1 | 0
ASPERGILLUS INFECTION (Infections and infestations) | 2 | 0
BACTERAEMIA (Infections and infestations) | 1 | 0
BACTERIAL INFECTION (Infections and infestations) | 1 | 0
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 1 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 1
DIABETIC GANGRENE (Infections and infestations) | 0 | 1
DIVERTICULITIS (Infections and infestations) | 2 | 0
ENDOCARDITIS (Infections and infestations) | 0 | 1
ESCHERICHIA INFECTION (Infections and infestations) | 1 | 0
FEBRILE INFECTION (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 2 | 2
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 0 | 1
GASTROENTERITIS SALMONELLA (Infections and infestations) | 1 | 0
GROIN INFECTION (Infections and infestations) | 0 | 1
H1N1 INFLUENZA (Infections and infestations) | 1 | 0
HERPES SIMPLEX (Infections and infestations) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 1 | 1
HERPES ZOSTER INFECTION NEUROLOGICAL (Infections and infestations) | 0 | 1
INFECTED LYMPHOCELE (Infections and infestations) | 0 | 1
INFECTION (Infections and infestations) | 3 | 1
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 1 | 0
INFLUENZA (Infections and infestations) | 0 | 1
OTITIS EXTERNA (Infections and infestations) | 0 | 1
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 2 | 0
PNEUMONIA (Infections and infestations) | 6 | 2
SEPTIC SHOCK (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0
TUBERCULOSIS (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
URETERITIS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
WOUND INFECTION (Infections and infestations) | 0 | 1
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 2 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
INFLAMMATORY MARKER INCREASED (Investigations) | 1 | 0
WEIGHT INCREASED (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PLASMACYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
MYOCLONIC EPILEPSY (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 2 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 | 1
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 2 | 0
HAEMATURIA (Renal and urinary disorders) | 1 | 0
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 2
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 | 0
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 1 | 0
MEDICAL DEVICE REMOVAL (Surgical and medical procedures) | 1 | 0
ANEURYSM (Vascular disorders) | 0 | 1
ANGIOPATHY (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 | 0
HYPERTENSION (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CNI-regimen (N=84) | CNI-free-regimen (N=78)
ANAEMIA (Blood and lymphatic system disorders) | 6 | 7
LEUKOPENIA (Blood and lymphatic system disorders) | 10 | 10
SINUS TACHYCARDIA (Cardiac disorders) | 3 | 5
TACHYCARDIA (Cardiac disorders) | 8 | 7
HYPERTHYROIDISM (Endocrine disorders) | 6 | 4
APHTHOUS ULCER (Gastrointestinal disorders) | 4 | 5
DIARRHOEA (Gastrointestinal disorders) | 11 | 5
NAUSEA (Gastrointestinal disorders) | 10 | 6
VOMITING (Gastrointestinal disorders) | 5 | 2
FATIGUE (General disorders) | 3 | 4
OEDEMA (General disorders) | 5 | 2
OEDEMA PERIPHERAL (General disorders) | 17 | 20
PYREXIA (General disorders) | 8 | 5
BRONCHITIS (Infections and infestations) | 8 | 3
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 11 | 4
NASOPHARYNGITIS (Infections and infestations) | 23 | 12
ORAL HERPES (Infections and infestations) | 2 | 5
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 4
BLOOD CREATININE INCREASED (Investigations) | 5 | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 5 | 3
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 7 | 3
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 9 | 5
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 8 | 6
HYPERURICAEMIA (Metabolism and nutrition disorders) | 5 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 7 | 13
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 7 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 | 1
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 2 | 5
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 1
HEADACHE (Nervous system disorders) | 5 | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 | 5
ACNE (Skin and subcutaneous tissue disorders) | 3 | 6
RASH (Skin and subcutaneous tissue disorders) | 5 | 2
HYPERTENSION (Vascular disorders) | 9 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-01-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT00862979/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT00862979/SAP_001.pdf